CLINICAL TRIAL: NCT03071835
Title: A Comparative Study of Subjects tHree to Thirteen Years Past thEiR fInal Follow-ON Visit. (Hyperion Study)
Brief Title: A Comparative Study of Subjects Past Their Final Follow-ON Visit
Acronym: HYPERION
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joshua M Hare, Louis Lemberg Professor of Medicine Director, Interdisciplinary Stem Cell Institute, University of Miami
Other Study IDs: 20150899
Record Dates: First submitted 2017-02-13; First posted 2017-03-07 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cardiomyopathies; Heart Diseases; Aging Frailty
Keywords: Stem Cells; Cardiovascular; Quality of Life; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Genetic testing will consist of collecting tissue and/or blood stored for future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A comparative study to follow subjects who received stem cell therapies three, five, seven, nine, and thirteen years after their follow-on visit. Subjects will be selected from a pool of previous Interdisciplinary Stem Cell Institute trial participants.

DETAILED DESCRIPTION:
A comparative study to follow subjects who received stem cell therapies three, five, seven, nine, and thirteen years after their follow-on visit. Subjects will be selected from a pool of previous Interdisciplinary Stem Cell Institute trial participants.

Subjects will be followed during the study depending on the initial visit for this trial. The time point at which they are followed will depend on the subject's injection date in the previous trial. Depending on the subjects first treatment date (Day of injection) in the previous Interdisciplinary Stem Cell Institute (ISCI) cardiovascular clinical trial, subjects may be eligible for one to four study visits in this trial. Those who do not have a three, five, seven, nine or eleven year visit may receive informed consent at the year thirteen visit. Thus, subjects can be enrolled and consented at any visit if the previous eligible visit was missed.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age and older
* Provide written informed consent
* Have been previously enrolled or currently participating in an investigator-initiated cardiovascular trial at ISCI (In cases where participants are currently enrolled in another clinical trial they are still able to participate concurrently in this trial).

Exclusion Criteria:

* Have known, serious radiographic contrast allergy, which cannot be managed with premedication only if able to undergo MRI or CT.
* Have a history of drug or alcohol abuse within the past 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study will consist of subjects who previously participated at an ISCI Trial and who are able to consent to being followed past their Follow-On visit.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Continued Improvement in subject's symptoms | at 3, 5, 7, 9, and 13 Years
  Demonstrate change of subject's symptoms by assessing cardiac events over an extended period of time following participation in an ISCI cardiac trial where the subject received Investigational product.

SECONDARY OUTCOMES:
Change in Cardiac Function via Cardiac MRI | at 3, 5, 7, 9, and 13 Years
  Evaluate Cardiac Function for changes, positive and negative via Cardiac MRI
Change in Cardiac Function via Cardiac CT | at 3, 5, 7, 9, and 13 Years
  Evaluate Cardiac Function for changes, positive and negative via Cardiac CT
Evaluate Functional Capacity via the NYHA Class | at 3, 5, 7, 9, and 13 Years
  Evaluate Functional Capacity via New York Heart Association (NYHA) Class Determination
Evaluate Functional Capacity via the Six Minute Walk Test | at 3, 5, 7, 9, and 13 Years
  Evaluate Functional Capacity via the Six Minute Walk Test
Evaluate change in Quality of Life via the Minnesota Living with Heart Failure | at 3, 5, 7, 9, and 13 Years
  Evaluate Quality Of Life Changes via Minnesota Living with Heart Failure (MLHF) Questionnaire
Evaluate change in Symptoms via cardiac events | at 3, 5, 7, 9, and 13 Years
  Evaluate Progression or Regression of disease (i.e. death, Left Ventricular Assist Device (LVAD), heart transplant and/or continuous intravenous infusion therapy (dobutamine, Milrinone, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, Md, Principal Investigator — University of Miami
Locations (1):
- ISCI / University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School of Medicine — http://isci.med.miami.edu